CLINICAL TRIAL: NCT04742348
Title: Research on Translational Outcomes of Alcohol (Project RETRO)
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: COVID-19 and expiration of funding
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Brittney Hultgren, Acting Assistant Professor Department of Psychiatry and Behavioral Sciences, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00009051
Record Dates: First submitted 2020-11-09; First posted 2021-02-08 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Alcohol Drinking
MeSH Terms: conditions — Alcohol Drinking | interventions — carbidopa, levodopa drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control, Placebo (Placebo Comparator): Similar looking tablet(s) to active drug will be administered in a single dose to those who are randomly assigned to this group.
  Interventions: Drug: Placebo
- Active Drug, Carbidopa + Levodopa (Experimental): Single dose of immediate release carbidopa-levodopa (50mg/500mg).
  Interventions: Drug: Carbidopa Levodopa

INTERVENTIONS:
Drug: Carbidopa Levodopa — Participants who are randomized to active drug group will receive 1 dose of immediate release carbidopa-levodopa (50mg/500mg) .
  Arms: Active Drug, Carbidopa + Levodopa
Drug: Placebo — Participants who are randomized to placebo group will be provided with similar looking tablet(s) as the active drug.
  Arms: Control, Placebo

SUMMARY:
The primary aim of the current study is to assess the effect of a single dose of carbidopa-levodopa on ad libitum alcohol consumption and alcohol craving in young adults with a history of binge drinking.

DETAILED DESCRIPTION:
This is a small (N = 42) 2-arm, double-blind, randomized controlled pilot study to assess the effect of a single dose of immediate release carbidopa-levodopa (50mg/500mg) to acutely reduce alcohol consumption and craving in college students with a history of heavy episodic drinking. Participants will be between 21-24 years old from 2- and 4- year colleges in the Seattle Metropolitan area. Interested students will contact the study line and provide verbal consent to be sent a link to an online screening survey. Eligible participants will be scheduled to come in for the ad libitum alcohol administration. Participants will receive either the carbidopa-levodopa or a placebo and complete the alcohol administration protocol.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in 2- or 4-year college program
* Currently living in the Seattle Metropolitan area
* Have at least two or more episodes of heavy episodic drinking (4/5 or more drinks in a 2 hours for women/men) in the past 30 days.

Exclusion Criteria:

* Exclusion criteria include:
* past-month severe alcohol or other substance use disorders,
* mood or anxiety disorder
* suicidal ideation
* risk of psychotic disorders
* excessive alcohol use reaching a Blood Alcohol Level greater than .30%
* history of serious medical conditions, regular use of prescription psychotropic or pain medication
* history of negative reactions to alcohol
* history of treatment for alcohol use disorder
* pregnancy or nursing.
* use of non-selective monoamine oxidase inhibitors in the past 2 weeks.
* narrow-angle glaucoma
* undiagnosed skin lesions,
* have a history of melanoma, cardiac issues or peptic ulcer.
* Currently taking or prescribed any form of levodopa or D2 agonists, D2 antagonists, isoniazid, methylphenidate, bupropion, Viagra, or phosphodiesterase inhibitors.

Ages: 21 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Alcohol Consumption | 1 hour
  Number of alcoholic drinks consumed
Alcohol Craving | 30 minutes in to alcohol administration
  Amount of alcohol craving as assessed by the Alcohol Urge Questionnaire by Bohn, Krahn & Staehler (1995)

SECONDARY OUTCOMES:
Alcohol craving | At the end of alcohol administration. Alcohol administration is 1 hour.
  Amount of alcohol craving as assessed by the Alcohol Urge Questionnaire by Bohn, Krahn & Staehler (1995)

CONTACTS AND LOCATIONS:
Overall Officials: Brittney Hultgren, PhD, Principal Investigator — University of Washington